CLINICAL TRIAL: NCT05357768
Title: Global collaboRAtion on CIC-DUX4, BCOR-CCN3, High-grade Undifferentiated Round Cell Sarcoma (URCS) Project
Acronym: GRACefUl
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: GRACefUl
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Undifferentiated Round Cell Sarcoma
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- retrospective cohort: Patients with undifferentiated round cell sarcomas treated from 01 January 1983 to April 2019 will be included.
  For retrospective analysis, it is expected to include about 200 patients.
  Interventions: Other: data collection and analysis on Formalin-fixed paraffin embedded tissue and/or frozen tumoral tissue
- prospective cohort: prospective patients with undifferentiated round cell sarcomas will be included in the study. For prospective study, it is expect to include 60 patients.
  Interventions: Other: data collection and analysis on Formalin-fixed paraffin embedded tissue and/or frozen tumoral tissue

INTERVENTIONS:
Other: data collection and analysis on Formalin-fixed paraffin embedded tissue and/or frozen tumoral tissue — Formalin-fixed paraffin embedded tissue and/or frozen tumoral tissue of cases negative for all Ewing's sarcoma molecular fusions, will be analyzed for the presence of CIC-DUX4 / BCOR-CCNB3 translocations fusion at each Institution.
  Treatment, outcome, and prognostic factors will be related with the molecular re-classification.

SUMMARY:
Experimental study with biological material : case series review of clinical and histological data

DETAILED DESCRIPTION:
This is a multicenter retrospective and prospective study that will analyze all cases with a diagnosis of Undifferentiated round cell sarcomas from 01 January 1983 and all new cases referring to each participant site.

ELIGIBILITY:
Inclusion Criteria:

* Patients with undifferentiated round cell sarcomas treated from 01 January 1983 and all new patients will be included.
* Clinical and outcome information available.
* Histological slides/formalin-fixed paraffin-embedded tissue tumor blocks from archive available to perform the histology analysis/frozen tissue representative of the tumor available.

Exclusion Criteria:

* Diagnosis different from undifferentiated round cell sarcomas
* Patient with no clinical or outcome information available

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: male and femalke patient without limit of age with a diagnosis of undifferentiated round cell sarcomas treated from 01 January 1983 and all new cases referring to each participant site.
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2019-06-11 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
event free survival | baseline
  Correlate clinical and pathological variables with event-free survival and overall-survival in undifferentiated round cell sarcomas.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCs Istituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/68/NCT05357768/Prot_001.pdf